CLINICAL TRIAL: NCT04164459
Title: A Multi-center, Randomized, Blinded Evaluator, Active Control, Parallel, Phase IV Study to Evaluate the Efficacy and Safety of Xalost S in Glaucoma Patients.
Brief Title: Evaluating the Efficacy and Safety of Xalost S in Glaucoma Patients.
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taejoon Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJO-002-401
Record Dates: First submitted 2019-10-15; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-09

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Xalost S (Experimental)
  Interventions: Drug: Xalost S
- Xalatan (Active Comparator)
  Interventions: Drug: Xalatan
- Taflotan-S (Active Comparator)
  Interventions: Drug: Taflotan-S

INTERVENTIONS:
Drug: Xalost S — One drop one times a day in study eye
  Arms: Xalost S
Drug: Xalatan — One drop one times a day in study eye
  Arms: Xalatan
Drug: Taflotan-S — One drop one times a day in study eye
  Arms: Taflotan-S

SUMMARY:
In patients with Glaucoma, Xalost S or Xalatan or Taflotan-S are administered for 12 weeks. After 12 weeks, among them, Xalatan administration group are switched to Xalost S or Taflotan-S. Extension study period is 8 weeks.

To compare effect (ocular surface damage) and safety of preservative-free Latanoprost/Tafluprost to Benzalkonium chloride-preserved Latanoprost in primary open angle glaucoma or normal tension glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female diagnosed with glaucoma, age 19 or over
* Written informed consent to participate in the trial

Exclusion Criteria:

* Patients who have received or have plans lacrimal puntual occulsion
* Use of contact lenses
* Any other Glaucoma except primary open angle glaucoma/normal tension glaucoma (ex) Closed anterior chamber angle/ angle-closure Glaucoma)
* Any condition limiting patient's ability to participate in the trial

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-12 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Corneal Staining Score at week 12 | week 12
  At week 12 of drug administration compare the therapeutic effectiveness between control drug and trial drug evaluated as the effect on corneal staining score.
  Scale: "Oxford grading system" that divides into 6 groups according to severity from 0 (absent) to 5 (severe).
  The higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Change from baseline in Hyperemia Score at week 4, 8, 12 | baseline and week 4, 8, 12
  After 4, 8, 12 weeks of drug administration compare the therapeutic effectiveness between control drug and trial drug evaluated as the effect on Hyperemia Score.
  Scale: "Efron Grading Scales" that divided into 5 groups according to severity from 0 (normal) to 4 (severe).
  The higher scores mean a worse outcome.
Change from baseline in Intraocular Pressure at week 4, 8, 12 | baseline and week 4, 8, 12
  After 4, 8, 12 weeks of drug administration compare the therapeutic effectiveness between control drug and trial drug evaluated as the effect on Intraocular pressure.
  The highest Intraocular pressure means a worse outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Taejoon Pharmaceutical Co., Ltd., Seoul, South Korea